CLINICAL TRIAL: NCT07343076
Title: Efficacy of Immediate Versus Staged Complete Revascularization in Patients With NSTE-ACS and Multivessel Disease (FUTURE II)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: People's Hospital of Xinjiang Uygur Autonomous Region (Other); LanZhou University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUTURE II
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: NSTEMI; NSTEMI - Non-ST Segment Elevation MI; Non-ST-elevation Acute Coronary Syndrome; NSTE-ACS (NSTEMI and UA)
Keywords: NSTEMI; FUTURE II
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Complete Revascularization (Experimental)
  Interventions: Device: Immediate Complete Revascularization
- Staged Complete Revascularization (Active Comparator)
  Interventions: Device: Staged Complete Revascularization

INTERVENTIONS:
Device: Immediate Complete Revascularization — Immediate Complete Revascularization: Emergency PCI for the culprit vessel is performed successfully, and simultaneous PCI is conducted for non-culprit vessels that meet the defined criteria (visually estimated diameter ≥2.5 mm, eligible for successful PCI, and visually estimated maximum diameter stenosis ≥ 70% or positive coronary physiology testing).
  Arms: Immediate Complete Revascularization
Device: Staged Complete Revascularization — During emergency intervention, PCI is performed only on the culprit vessel. Elective PCI is then conducted for non-culprit vessels that meet the defined criteria (visually estimated diameter ≥ 2.5 mm, eligible for successful PCI, and visually estimated maximum diameter stenosis ≥ 70% or positive coronary physiology testing)-either during the current emergency hospitalization or within 6 weeks after the culprit vessel PCI.
  Arms: Staged Complete Revascularization

SUMMARY:
This is a prospective, multi-center, randomized controlled, open-label, blinded endpoint assessment study. The objective is to compare the 1-year incidence of major adverse cardiovascular and cerebrovascular events (MACCE) between two treatment strategies-immediate complete revascularization and staged complete revascularization-in NSTE-ACS patients with multivessel disease (MVD).

NSTE-ACS patients who meet other the inclusion and exclusion criteria will be randomized into the following two groups after signing an informed consent form:

Intervention group Immediate Complete Revascularization: Emergency PCI for the culprit vessel is performed successfully, and simultaneous PCI is conducted for non-culprit vessels that meet the defined criteria (visually estimated diameter ≥2.5 mm, eligible for successful PCI, and visually estimated maximum diameter stenosis ≥ 70% or positive coronary physiology testing).

Control group During emergency intervention, PCI is performed only on the culprit vessel. Elective PCI is then conducted for non-culprit vessels that meet the defined criteria (visually estimated diameter ≥ 2.5 mm, eligible for successful PCI, and visually estimated maximum diameter stenosis ≥ 70% or positive coronary physiology testing)-either during the current emergency hospitalization or within 6 weeks after the culprit vessel PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years or older.
2. Patients with intermediate-to-high risk NSTE-ACS who meet the diagnostic criteria specified in current guideline, complicated by multivessel coronary artery disease, and have successfully undergone PCI for the culprit vessel.
3. PCI within 72 hours of diagnosis.
4. Accompanied by multivessel disease: defined as at least one non-culprit artery that meets the following conditions: a diameter of ≥2.5 mm by visual inspection, which can be successfully subjected to PCI, and the most severe diameter stenosis rate by visual inspection is at least 70% or positive coronary physiology testing.
5. Sign an informed consent form before participating in the study.

Exclusion Criteria:

1. Have received thrombolytic treatment.
2. Cardiogenic shock or SBP< 90 mmHg.
3. Patients in whom the culprit vessel cannot be clearly identified.
4. Left main coronary artery lesion, non-infarct-related arteries are CTO lesions or severely calcified lesions, complex lesions that require the use of special devices such as rotational ablation/laser.
5. Previous PCI within the past 1 month or previous coronary artery bypass graft (CABG).
6. Accompanied by other diseases that lead to an expected survival time of ≤ 12 months.
7. Patients with other serious diseases such as severe renal insufficiency (creatinine clearance value <30ml/min), hepatic insufficiency, thrombocytopenia (≤50*109/L).
8. Patients with severe valvular disease, hypertrophic cardiomyopathy, restrictive cardiomyopathy, and primary pulmonary hypertension.
9. Not suitable for clinical study:

   1. Have enrolled in the other clinical studies that may affect the outcome assessment of this study.
   2. Pregnant and lactating women.
   3. Known allergy to the drugs that may be used in the study.
   4. Unable to comply with the trial protocol or follow-up requirements; or the investigator believes that participation in the trial may put the patient at greater risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1904 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular event (MACCE) | at 1 year after randomization
  defined as a composite of all-cause death, non-fatal myocardial infarction, unplanned ischemia-driven revascularization, and stroke

SECONDARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular event (MACCE) | 1 month, 6 months, 2 years, 3 years after randomization
  defined as a composite of all-cause death, non-fatal myocardial infarction, unplanned ischemia-driven revascularization, and stroke
All-cause death | 1 month, 6 months, 1 year, 2 years, 3 years after randomization
  cardiovascular, non-cardiovascular, death of undetermined cause
Cardiac death | 1 month, 6 months, 1 year, 2 years, 3 years after randomization
Myocardial infarction | 1 month, 6 months, 1 year, 2 years, 3 years after randomization
  target vessel related, non-target vessel related
Target vessel revascularization | 1 month, 6 months, 1 year, 2 years, 3 years after randomization
  ischemia-driven, non-ischemia-driven
Any coronary revascularization | 1 month, 6 months, 1 year, 2 years, 3 years after randomization
  ischemia-driven, non-ischemia-driven
ARC-2 defined stent thrombosis | 1 month, 6 months, 1 year, 2 years, 3 years after randomization
  including confirmed and possible stent thrombosis in acute, subacute, and late time frames
Stroke | 1 month, 6 months, 1 year, 2 years, 3 years after randomization
  ischaemia, hemorrhage
Contrast agent-related acute kidney injury | 1 month after randomization
Major bleeding | 1 month, 6 months, 1 year, 2 years, 3 years after randomization
  BARC grades 3 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, MD, PhD, Principal Investigator — RenJi Hospital; Yining Yang, MD, PhD, Principal Investigator — People's Hospital of Xinjiang Uygur Autonomous Region; Ming Bai, MD, PhD, Principal Investigator — LanZhou University

IPD SHARING:
Plan to Share IPD: Yes
Bona fide researchers can request access to the data after the publication of the main results, provided that a study protocol is submitted to and approved by the FUTURE II Steering Committee.
Supporting Information: Study Protocol, SAP
Time Frame: Data sharing will be available from 12 months after the publication of the main results.
Access Criteria: 1. The data sharing will be only for the purposes of health and medical research and within the constraints of the consent under which the data were originally gathered.
  2. The Custodian of the Collection will not consider any Proposals for data sharing that unblind, or potentially unblind, randomised comparisons in active / ongoing trials.
  3. Requesters should be employees of a recognised academic institution, health service organisation, commercial research organisation or from the pharmaceutical industry. Requesters must have experience in medical research.
  4. Requesters must be able to demonstrate through their peer review publications in the area of interest their ability to carry out the proposed use of the requested dataset from a Collection.
  5. The Requesters must not have a conflict of interest that may potentially influence their interpretation of any analyses.